CLINICAL TRIAL: NCT07272707
Title: Psychometric Hepatic Encephalopathy Score in Prediction of Minimal Hepatic Encephalopathy in Compensated Cirrhotic Patients
Acronym: PHES-MHE
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Sabry Thabit, Sohag , Akhmim, Schools street, Sohag University
Other Study IDs: Soh-Med--25-11-9MS
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Minimal Hepatic Encephalopathy
Keywords: Minimal hepatic encephalopathy; Psychometric Hepatic Encephalopathy Score

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Cirrhotic Patients (Cases): Compensated cirrhotic patients aged 18-70 years undergoing Psychometric hepatic encephalopathy score testing.
  Interventions: Other: Psychometric Hepatic Encephalopathy Score (PHES)
- Group 2: Healthy Volunteers (Controls): Healthy adults aged 18-70 years with no chronic disease and normal cognitive function undergoing Psychometric hepatic encephalopathy score testing.
  Interventions: Other: Psychometric Hepatic Encephalopathy Score (PHES)

INTERVENTIONS:
Other: Psychometric Hepatic Encephalopathy Score (PHES) — A standardized paper-and-pencil neuropsychological test battery used to detect minimal hepatic encephalopathy. It includes:
  1. Number Connection Test A (NCT-A)
  2. Number Connection Test B (NCT-B)
  3. Digit Symbol Test (DST)
  4. Serial Dotting Test (SDT)
  5. Line Tracing Test (LTT)
  Tests are administered in a quiet environment between 8 AM and 3 PM by trained personnel. Performance is recorded as completion time, error score, or point score depending on test type.

SUMMARY:
Minimal hepatic encephalopathy (MHE) is a covert form of hepatic encephalopathy associated with cognitive and psychomotor impairment in patients with compensated liver cirrhosis. Early detection of MHE is crucial to prevent progression to overt encephalopathy. The Psychometric Hepatic Encephalopathy Score (PHES) is a validated neuropsychological test battery for diagnosing MHE. This study aims to screen for MHE among compensated cirrhotic patients using PHES and to compare performance with healthy matched controls.

DETAILED DESCRIPTION:
This cross-sectional case-control study will include compensated cirrhotic patients aged 18-70 years attending Sohag University Hospital, as well as a control group of healthy volunteers matched for age and education. All participants will undergo clinical evaluation, laboratory investigations, abdominal ultrasound, and psychometric assessment using the PHES battery (NCT-A, NCT-B, DST, SDT, LTT). PHES performance will be compared between cases and controls. The diagnostic accuracy of PHES for detecting MHE will be evaluated using sensitivity, specificity, PPV, NPV, and AUROC. Correlation analyses will explore associations between PHES scores and liver disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria (Cirrhotic Patients):

  1. Age 18-70 years.
  2. Diagnosed compensated liver cirrhosis, regardless of etiology.
  3. Able to read and write.
  4. Adequate vision, hearing, and physical ability to perform the PHES tests.

     Inclusion Criteria (Healthy Controls):

  <!-- -->

  1. Age 18-70 years.
  2. No chronic medical, neurological, psychiatric, renal, or cardiac disease.
  3. Able to read and write.
  4. Adequate cognition, hearing, vision, and physical ability.

     Exclusion Criteria:

  <!-- -->

  1. Chronic liver disease.
  2. Neuropsychiatric illness.
  3. Use of psychoactive medications.
  4. Illiteracy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Cirrhotic Patients (Cases)
  Compensated cirrhotic patients aged 18-70 years undergoing PHES testing.
  Group 2: Healthy Volunteers (Controls)
  Healthy adults aged 18-70 years with no chronic disease and normal cognitive function.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate of minimal hepatic encephalopathy using PHES | Baseline assessment
  Proportion of compensated cirrhotic patients classified as having minimal hepatic encephalopathy based on PHES total score and normative regression equations.

SECONDARY OUTCOMES:
Comparison of PHES subtest performance between cirrhotic patients and healthy controls | Baseline
  Differences in NCT-A, NCT-B, DST, SDT, and LTT scores between groups.
Association between PHES total score and liver disease severity | Baseline
  Correlation of PHES with Child-Pugh score, ALT, AST, albumin, bilirubin, INR.

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available upon reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication of study results.
Access Criteria: Data may be shared with investigators who submit a justified request via email.